CLINICAL TRIAL: NCT07153237
Title: A Prospective, Multicentric, Randomized, Evaluator-blind, Controlled, Interventional Clinical Investigation Evaluating the Clinical Performance and Safety of STYLAGE® HydroMax, a Hyaluronic Acid-based Gel
Brief Title: Clinical Performance and Safety of STYLAGE® HydroMax
Acronym: FHAME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Collaborators: Quantificare SA (Unknown); Eurofins Dermscan Pharmascan (Industry); Inferential (Industry); International Clinical Trials Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIV-STYL-HYDM-02; 2025-A00467-42 (Other: ANSM)
Record Dates: First submitted 2025-08-21; First posted 2025-09-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Aging; Aesthetic
Keywords: Hyaluronic Acid; Aging; Aesthetics; Healthy subjects; Injection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention Arm (Group A): two injection sessions with STYLAGE® HydroMax before Week 6 (Experimental): Subjects will be randomized 2:1 to Group A. During Stage 1, they will receive two STYLAGE® HydroMax injection sessions at baseline and Week 3. In Stage 2, they will be followed for 30 additional weeks (up to Week 36) and will receive a third injection at Week 24 after the first injection.
  Interventions: Device: STYLAGE® HydroMax
- Control Arm (Group B): No Treatment before Week 6 (Other): Subjects will be randomized 2:1 to Group B. In Stage 1, they will receive no treatment until Week 6. Data collected at Week 6 will serve as pre-treatment baseline. In Stage 2, eligible subjects in Group B will receive STYLAGE® HydroMax following the same schedule as Group A. All subjects in Group B will be followed up to 36 weeks after their first STYLAGE® HydroMax injection.
  Interventions: Device: STYLAGE® HydroMax

INTERVENTIONS:
Device: STYLAGE® HydroMax — 3 injection sessions : Group A: at week 0 (V1a), week 3 (V2a), and week 24 (V5a). Group B: at week 6 (V3b), week 3 from V3b (V4b), and week 24 from V3b (V7b)

SUMMARY:
FHAME is a post-market clinical investigation designed to strengthen the clinical evidence supporting the effectiveness of STYLAGE® HydroMax in the treatment of superficial wrinkles, primarily on the cheeks.

DETAILED DESCRIPTION:
FHAME is an interventional, post-market, multicentric, prospective, randomized clinical investigation conducted in subjects without any pathology, treated with CE-marked STYLAGE® HydroMax to confirm and update its clinical performance and safety. The primary objective of the study is to assess the mean change from baseline in cheek wrinkle severity, evaluated by an independent blinded assessor at six weeks post-baseline using the Bazin cheek wrinkle scale during live assessments. Clinical performance will be demonstrated if the mean change in the Bazin cheek wrinkle score at six weeks post-baseline is statistically superior in the treatment group (Group A) compared to the control group (Group B). To demonstrate the superiority of STYLAGE® HydroMax compared to no treatment, a total of 81 subjects will be randomized in the study. The overall duration of the study is expected to be approximately seventeen months, including a recruitment period of around six months, a screening period of two weeks, and an investigation period of thirty-six weeks post-randomization for Group A and forty-two weeks for Group B.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects without any pathology aged between 35 and 70 years old at inclusion.
2. Subjects wishing treatment for the aesthetic improvement of facial wrinkles.
3. Subject having given freely and expressly their informed consent.
4. Subject with a Grade 2 to 5 score on the Bazin cheek wrinkle scale.
5. Subject with the same wrinkle score according to the Bazin cheek wrinkle scale for both cheeks (i.e., symmetrical cheeks).
6. Subject psychologically able to understand investigation related information and to give written informed consent.
7. Subject affiliated to a health social security system.
8. Female of childbearing potential must use a medically accepted contraceptive regimen for at least 12 weeks prior to the start of the investigation and for the duration of the investigation.
9. Subject agreeing not to change any hormonal treatment (including contraceptive treatment and hormone replacement therapy) for the duration of the investigation.
10. Subject agreeing to keep their usual cleansing / care products for the duration of the investigation.
11. Subject agreeing to apply a SPF50 cream when exposed to non-intensive sunlight (i.e., excluding prolonged sun exposure such as sunbathing or extended beach exposure).
12. Subject able to comply with investigation requirements and complete all required visits.
13. Subject agreeing not to receive any other plastic surgery or cosmetic procedure on the face (e.g. dermal fillers, toxin-based treatment, fractional or ablative laser, micro-dermabrasion, chemical peel, noninvasive procedures for skin laxity) for the duration of the investigation.
14. Subject agreeing not to have any planned dental surgery during the investigation.

Exclusion Criteria:

1. Pregnant or breastfeeding woman or woman planning a pregnancy during the investigation.
2. Woman less than a year past menopause.
3. Subject with a tattoo, a scar, moles, too many hairs or body hairs (i.e. beard), or anything on the studied zones which might interfere with outcome evaluations.
4. Subject who has been deprived of their freedom by administrative or legal decision or who is under guardianship.
5. Member of the investigating team or family member of a member of the investigating team.
6. Subject in a social or sanitary establishment.
7. Subject having received 6000 euros indemnities for participation in research involving human beings in the 12 previous months, including participation in the present investigation.
8. Subject participating in another research on human beings or who is in an exclusion period of one.
9. Subject who had intensive exposure to sunlight (i.e., prolonged sun exposure such as sunbathing or extended beach exposure) or UV-rays within the previous month and/or for whom intensive exposure to sunlight or UV-rays is foreseen during the clinical investigation.
10. Subject suffering from severe or progressive disease or any other pathology that may interfere with the evaluation of the investigation results.
11. Subject with known history of, or suffering from, autoimmune disease and/or immune deficiency.
12. Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…). Subject with recurrent herpes in the midface area is eligible if asymptomatic at time of inclusion.
13. Subject having a history of severe allergy or anaphylactic shock including hypersensitivity to HA or to one of the components of the tested device, to antiseptic solution or anesthesia products if applicable.
14. Subject with a history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats.
15. Subject predisposed to keloids or hypertrophic scarring.
16. Subject prone to develop inflammatory skin conditions or has a tendency to bleeding disorders.
17. Subject with a fructose intolerance.
18. Subject who had dental surgery within the 6 weeks prior to the start of the investigation.
19. Subject having received treatment with laser, dermabrasion, surgery, deep chemical peeling, or other ablative procedure on the investigated areas within the 12 months prior to start of the investigation.
20. Subject having received injections of botulinum toxin within the 9 months prior to the start of the investigation.
21. Subject having received an injection with a resorbable filling product in the investigated areas within the 18 months prior to the start of the investigation.
22. Subject having previously received at any time in the past 24 months an injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of HA and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate…) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles …).
23. Subject having previously received at any time in the past 24 months a treatment with tensor threads on the face.
24. Subject having taken medication such as aspirin, non-steroidal anti-inflammatory drugs (NSAIDs) (ibuprofen, naproxen…), antiplatelet agents, anticoagulants, vitamin C in the week prior each injection session or who is a chronic user of these medications.
25. Subject undergoing a topical treatment on the test areas or taking either of the following systemic treatments:

    1. Antihistamines within the 2 weeks prior to the start of the investigation.
    2. Immunosuppressors and/or corticoids within the 4 weeks prior to the start of the investigation.
    3. Retinoids within the 6 months prior to the start of the investigation

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Mean changes in cheek wrinkle score (independant blinded evaluator) | 6 weeks port-baseline
  Mean change from baseline in cheek wrinkle severity score assessed by an independent blinded evaluator at 6 weeks (V3a/V3b) post-baseline using the 8-grade Bazin cheek wrinkle scale (0 = no wrinkles, 8 = most severe wrinkles) during live assessments.

SECONDARY OUTCOMES:
Mean changes in cheek wrinkle score (live assessments) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in cheek wrinkle score assessed using the 8-grade Bazin cheek wrinkle scale (0 = no wrinkles, 8 = most severe wrinkles) during live assessments:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no-treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis.
Percentages of improved subjects in cheek wrinkle score (live assessments) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Percentages of improved subjects, assessed using the 8-grade Bazin cheek wrinkle scale (0 = no wrinkles, 8 = most severe wrinkles) during live assessments:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no-treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis.
Mean changes in cheek wrinkle score (central review) | From baseline to 3 post-baseline and from pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in cheek wrinkle score assessed using the 8-grade Bazin cheek wrinkle scale (0 = no wrinkles, 8 = most severe wrinkles) by central review: From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b). From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment.
Percentages of improved subjects in cheek wrinkle score (central review) | From baseline to 3 and 6 weeks post-baseline. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement.
  Percentages of improved subjects, assessed using the 8-grade Bazin cheek wrinkle scale (0 = no wrinkles, 8 = most severe wrinkles) by central review:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment.
Mean changes in crow's feet wrinkle score (live assessments) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in crow's feet wrinkle score assessed using the 6-grade Bazin crow's feet wrinkle scale (0 = no wrinkles, 6 = most severe wrinkles) during live assessments:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no-treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis
Percentages of improved subjects in crow's feet wrinkle score (live assessments) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Percentages of improved subjects, assessed using the 6-grade Bazin crow's feet wrinkle scale (0 = no wrinkles, 6 = most severe wrinkles) during live assessments:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no-treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis
Mean changes in crow's feet wrinkle score (central review) | From baseline to 3 and 6 weeks post-baseline. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement
  Mean changes in crow's feet wrinkle score assessed using the 6-grade Bazin crow's feet wrinkle scale (0 = no wrinkles, 6 = most severe wrinkles) by central review:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment
Percentages of improved subjects in crow's feet wrinkle score (central review) | From baseline to 3 and 6 weeks post-baseline. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement
  Percentages of improved subjects, assessed using the 6-grade Bazin crow's feet wrinkle scale (0 = no wrinkles, 6 = most severe wrinkles) by central review:
  From baseline (V1a/V1b) to 3 weeks post-baseline (V2a/V2b and 6 weeks (V3a/V3b) post-baseline.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment.
Mean changes in cheek and crow's feet wrinkle volume (3D photography) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in cheek and crow's feet wrinkle volume determined by central analysis of 3D photography:
  From baseline (V0 or V1a/V0 or V1b) to 3 weeks (V2a/V2b) and 6 weeks post-baseline (V3a/V3b), for the "no-treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis
Mean changes in cheek and crow's feet wrinkle depth (3D photography) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in cheek and crow's feet wrinkle depth determined by central analysis of 3D photography: From baseline (V0 or V1a/V0 or V1b) to 3 weeks (V2a/V2b) and 6 weeks post-baseline (V3a/V3b), for the "no-treatment" controlled stage analysis. From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis
Mean changes in cutaneous roughness of the crow's feet and cheek (3D photography) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in cutaneous roughness of the crow's feet and cheek areas determined by central analysis of 3D photography:
  * From baseline (V0 or V1a/V0 or V1b) to 3 weeks (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no-treatment" controlled stage analysis.
  * From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis.
Mean changes in cutaneous tension of the crow's feet and cheek (3D photography) | From pre-treatment baseline to 6 and 36 weeks post treatment
  Mean changes in cutaneous tension of the crow's feet and cheek areas determined by central analysis of 3D photography:
  From pre-treatment baseline (V0 or V1a/V3b) to 6 weeks (V3a/V5b), and 36 weeks (V6a/V8b) post treatment, for the final analysis.
Mean changes in skin thickness of the crow's feet and cheek (DermaScan C USB) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in skin thickness of the crow's feet and cheek areas determined using DermaScan C USB, a high frequency skin ultrasound used to visualize layers of the skin and subcutaneous tissues and to make approximate dimensional measurements:
  From baseline (V1a/V1b) to 3 weeks (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis
Mean changes in density of the crow's feet and cheek (DermaScan C USB) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in density of the crow's feet and cheek areas determined using DermaScan C USB, a high frequency skin ultrasound used to visualize layers of the skin and subcutaneous tissues and to make approximate dimensional measurements: From baseline (V1a/V1b) to 3 weeks (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no treatment" controlled stage analysis. From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis
Percentages of GAIS responders, assessed by the subject and the Evaluator | At 3, 6, 12, 24 and 36 weeks post-treatement
  Percentages of GAIS (Global Aesthetic Improvement Scale, rated on a 5-point scale) responders, assessed by the subject and the Evaluator:
  At 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post-treatment
Mean changes in subject's satisfaction scores for cheeks and crow's feet (FACE-Q) | From baseline to 3 and 6 weeks post-baseline for the "no-treatment" controlled stage analysis. From pre-treatment baseline to 3, 6, 12, 24 and 36 weeks post-treatement for the final analysis
  Mean changes in subject's satisfaction scores for cheeks and crow's feet treatment using the FACE-Q TM "Satisfaction with Skin", FACE-QTM "Satisfaction with Cheeks", FACE-QTM"Appraisal of Lines: Crow's feet", and FACE-QTM "Patient perceived age visual analogue scale" questionnaires (Rasch transformed score):
  From baseline (V1a/V1b) to 3 weeks (V2a/V2b) and 6 weeks (V3a/V3b) post-baseline, for the "no treatment" controlled stage analysis.
  From pre-treatment baseline (V1a/V3b) to subsequent visits at 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post treatment, for the final analysis.
Percentages of subjects who are satisfied and percentages of subjects for whom the Evaluator is satisfied for each item (satisfaction questionnaire) | At 3, 6, 12, 24 and 36 weeks post-treatement
  Percentages of subjects who are satisfied and percentages of subjects for whom the Evaluator is satisfied for each item of the satisfaction questionnaire (6-point sale):
  At 3 weeks (V2a/V4b), 6 weeks (V3a/V5b), 12 weeks (V4a/V6b), 24 weeks (V5a/V7b), and 36 weeks (V6a/V8b) post-treatment.
Mean pain scores during injection assessed by subject (10-cm visual analogue scale) | First injection session (V1a/V3b), the second injection session (V2a/V4b) and the third injection session (V5a/V7b)
  Mean pain scores during injection assessed by subject using a 10-cm visual analogue scale (VAS) ranging from 0 ("no pain at all") to 10 ("unbearable pain"):
  Within 5 minutes of the injections performed at the first injection session (V1a/V3b), the second injection session (V2a/V4b) and the third injection session (V5a/V7b)
Percentages of subjects for whom the Treating Investigators are satisfied of the usability of the device | First injection session (V1a/V3b), the second injection session (V2a/V4b) and the third injection session (V5a/V7b).
  Percentages of subjects for whom the Treating Investigators are satisfied with the usability of the device for each item of the questionnaire, assessed using six 10-point scale questions evaluating the usability of the HA gel in each area:
  Within 10 minutes after performing the injections at the first injection session (V1a/V3b), the second injection session (V2a/V4b) and the third injection session (V5a/V7b).
Percentages of subjects for whom the Treating Investigators are satisfied with the ease of massaging | First injection session (V1a/V3b), the second injection session (V2a/V4b) and the third injection session (V5a/V7b).
  Percentages of subjects for whom the Treating Investigators are satisfied with the ease of massaging, assessed using a 5-point scale for each area of the HA gel:
  Within 10 minutes after performing the injections at the first injection session (V1a/V3b), the second injection session (V2a/V4b) and the third injection session (V5a/V7b).
Occurrence of Injection Site Reactions (ISRs) to Assess Product Safety and Tolerability | Throughout the investigation period: V0, V1a/V1b, V2a/V2b, V3a/V3b, V4a/V4b, V5a/V5b, V6a/V6b, V7b, V8b
  Product safety and tolerance will be assessed by collection of the occurence of any Injection site reactions (ISRs).
  The following events occurring within 14 days after an injection session will be considered as ISR: redness/erythema, pain/tenderness, burning sensation, firmness/induration, sensitivity disorder, swelling/edema, lumps/bumps, bruising/ecchymosis with potential bleeding and hematoma, itching.
  An ISR can be requalified as an adverse event (AE) if, at the discretion of the principal investigator, the nature of the observation/event exceeds what would be expected and considered normal.
Occurrence of Adverse Events (AE) to Assess Product Safety and Tolerability | Throughout the investigation period: V0, V1a/V1b, V2a/V2b, V3a/V3b, V4a/V4b, V5a/V5b, V6a/V6b, V7b, V8b
  Product safety and tolerance will be assessed by collection of the occurence of any Adverse Events (AE).
  Any other events occurring at any time or any ISR (Injection Site Reaction) persisting beyond 14 days after an injection session will be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia MOREL-MANDRINO, MD, Principal Investigator — Eurofins Dermscan, Villeurbanne, FRANCE
Locations (2):
- France (2):
  - Eurofins DERMSCAN, Aix-en-Provence
  - Eurofins DERMSCAN PHARMASCAN, Villeurbanne

IPD SHARING:
Plan to Share IPD: No